CLINICAL TRIAL: NCT01414452
Title: Reperfusion Injury and Cardiac Remodelling After Myocardial Infarction in Relation to Adiponectin Level, Circulating Endothelial Progenitor Cells and Endothelial Microparticles
Brief Title: Role of Adiponectin and Endothelial Progenitor Cells in Reperfusion Injury in Patients With Acute Myocardial Infarction
Acronym: R²ACE
Status: Completed | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, M Claeys, Prof dr, Universiteit Antwerpen
Other Study IDs: UAntwerpen
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Myocardial Infarction; Reperfusion Injury
Keywords: Myocardial Infarction; Reperfusion injury; Adiponectin; endothelial progenitor cells
MeSH Terms: conditions — Myocardial Infarction; Reperfusion Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- STEMI patients: Patients with ST elevation myocardial infarction,lasting <12 hour, who were succesfully treated with primary PCI

SUMMARY:
There is experimental evidence that low levels of adiponectin are associated with more reperfusion injury. In addition experimental studies have demonstrated that endothelial progenitor cells may have a favorable effect on remodeling, mainly through stimulation of neo-revascularisation. Clinical data on these issues are lacking. This clinical project studies the role of adiponectin, endothelial progenitor cells and endothelial microparticles in the ischaemia-reperfusion process and the compensatory ventricular remodelling in a population of 250 infarction patients treated with primary PCI. If the role of these factors could be confirmed in this clinical setting, those factors might represent a new target for therapeutic interventions in AMI patients.

ELIGIBILITY:
Inclusion Criteria:

* STEMI treated with primary PCI

Exclusion Criteria:

* ischemia time >12h
* use of immunosuppressive therapy
* unsuccessful recanalisation
* not-interpretable ST-T segment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ST elevetion myocardial infarction patients
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
occurrence of reperfusion injury after succesfull primary PCI | within 90 min after PCI
  Serial ECG measurements (before and after PCI to assess extent of ST segment resolution as marker of reperfusion injury

SECONDARY OUTCOMES:
Major cardiovascular event rate | at 1 year
  combined endpoint of hospitalisation (or extension of hospitalisation) for heart failure and cardiac death in a period of one year

CONTACTS AND LOCATIONS:
Overall Officials: Marc Claeys, MD PHD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University hospital, Edegem, Antwerp, Belgium